CLINICAL TRIAL: NCT03732859
Title: A Prospective Observational Registry to Describe the Disease Course and Outcomes of Idiopathic Pulmonary Fibrosis Patients in a Real-world Clinical Setting. PROOF-Registry New and Extended Belgium -Luxembourg
Brief Title: PROOF-Registry New and Extended Belgium -Luxembourg
Acronym: PROOF-NEXT
Status: Completed | Type: Observational
Sponsor: Belgian Thoracic Society (Other)
Collaborators: Boehringer Ingelheim (Industry); Roche Farma, S.A (Industry)
Responsible Party: Sponsor
Other Study IDs: BVPSBP01
Record Dates: First submitted 2018-07-26; First posted 2018-11-07 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: IPF
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A Prospective Observational Registry to describe the disease course and outcomes of Idiopathic Pulmonary Fibrosis patients in a real-world clinical setting.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is a chronic disease of unknown etiology, characterized by scar tissue (fibrosis) within the lungs. IPF is one of the most common forms of interstitial lung disease and is associated with substantial morbidity and mortality (average survival of approximately three years from the time of diagnosis)).

The epidemiology and natural history of IPF is still not completely understood. Incidence and prevalence of IPF are difficult to determine because uniform diagnostic criteria have only recently been defined. Recent data among subjects aged 50 years or older suggests an age- and sex-adjusted incidence rate ranging from 8.8 cases to 17.4 cases per 100,000 person-years in the USA. In the same population, age- and sex- adjusted prevalence ranged from 27.9 cases to 63 cases per 100,000 persons.

Familial form of IPF accounts for 0.5 to 2% of all cases of IPF. Several environmental or occupational exposures seem to be prevalent in the medical histories of patients diagnosed with the disease.

The onset of IPF symptoms is slow, but symptoms become progressively worse over time. Breathlessness upon exertion and chronic dry cough are the major symptoms. Gastro-esophageal acid reflux is present in almost 90% of patients with IPF but often occurs without symptoms.

Auscultation of the lungs reveals early inspiratory crackles, predominantly located in the lower posterior lung zones upon physical exam. Clubbing is found in approximately 50% of patients with IPF.

Quality of life of patients with IPF is impacted by the disease.

Establishing an accurate diagnosis for the patient who presents with interstitial lung disease is an essential component of management. The recent ATS/ERS/JRS/ALAT recommendations on the diagnosis and management of IPF were developed from a systematic review of the published literature. High-resolution computed tomography (HRCT) scanning has a central role in the IPF diagnostic pathway with formal designation of criteria for an HRCT pattern of Usual Interstitial Pneumonia (UIP). In the correct clinical context, a UIP pattern on HRCT is indicative of a definite diagnosis of IPF without the need for a surgical lung biopsy.

IPF presents significant associations with other cardiopulmonary disorders including coronary artery disease, pulmonary embolism, sleep apnea, respiratory infections and lung cancer. In addition, patients with IPF are at risk for 'acute exacerbations'. Acute exacerbation is defined as an acute, clinically significant respiratory deterioration characterized by evidence of new widespread alveolar abnormality. Diagnostic criteria are: previous or concurrent diagnosis of IPF; acute worsening or development of dyspnea typically < 1 mo duration; computed tomography with new bilateral ground-glass opacity and/or consolidation superimposed on a background pattern consistent with usual interstitial pneumonia pattern; deterioration not fully explained by cardiac failure or fluid overload. These acute exacerbations are responsible for 50% of deaths in IPF and may affect previously stable patients.

The clinical course of IPF is highly variable and as a result, therapeutic strategies should be highly individualized, based upon the specific patients' medical history and co-morbidities.

Pirfenidone and Nintedanib are drugs approved for the treatment of adult patients with mild to moderate idiopathic pulmonary fibrosis in the European Union. In order to complement the data collected in previous studies, we implement a registry to describe the epidemiology and natural history of IPF, as well as the quality of life of IPF patients, and use of health care resources, in Belgium and Luxembourg. This registry will also enable the collection of clinical data of patients treated with Pirfenidone or Nintedanib and other therapies used in the treatment of IPF. The registry will be implemented in collaboration with pulmonologists and expert centers in order to enable the inclusion and follow up of recently diagnosed IPF patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* IPF diagnosis "definite" or "probable" (2011 ATS/ERS guidelines definitions) confirmed by a multidisciplinary team (= minimum of pulmonologist, radiologist, pathologist, all with expertise in IPF).
* Patients who agreed to participate in the registry and have completed and signed the Informed Consent Form

Exclusion Criteria:

* Patients incapable of giving informed consent
* Patients participating in a clinical trial at the time of inclusion in the registry and whose protocol does not allow participation in another trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with an IPF diagnosis "definite" or "probable" (according to 2011 ATS/ERS guidelines definitions) which is confirmed by a multidisciplinary team (= minimum of pulmonologist, radiologist, pathologist, all with expertise in IPF).
Sampling Method: Probability Sample
Enrollment: 575 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-01-09 (Actual)

PRIMARY OUTCOMES:
The first occurrence of a decrease of ≥ 10% in percent predicted forced vital capacity (FVC) since baseline. | overall duration of study (5 years)
  FVC data will be retrieved from the medical file of the participant.
The first occurrence of a decrease of ≥ 15% in percent predicted diffusing capacity of the lung for carbon monoxide (DLCO) since baseline | overall duration of study (5 years)
  DLCO data will be retrieved from the medical file of the participant.
Number of participants alive | overall duration of study (5 years)
  Data on death will be retrieved from the medical file of the participant.
The evolution of percent predicted forced vital capacity (FVC) | overall duration of study (5 years)
  FVC data will be retrieved from the medical file of the participant.
The evolution of percent predicted diffusing capacity of the lung for carbon monoxide (DLCO) | overall duration of study (5 years)
  DLCO data will be retrieved from the medical file of the participant.
The number of acute exacerbations of IPF | overall duration of study (5 years)
  Acute exacerbations of IPF data will be retrieved from the medical file of the participant.

SECONDARY OUTCOMES:
The number of patients per IPF treatment drug | overall duration of study (5 years)
  IPF treatment drug data will be retrieved from the medical file of the participant.
The mean initial dose per IPF treatment drug | overall duration of study (5 years)
  IPF treatment drug data will be retrieved from the medical file of the participant.
The mean number of dose changes per IPF treatment drug | overall duration of study (5 years)
  IPF treatment drug data will be retrieved from the medical file of the participant.
The number of participants who have discontinued the IPF treatment per IPF treatment drug | overall duration of study (5 years)
  IPF treatment drug data will be retrieved from the medical file of the participant.
The mean duration of treatment in days per IPF treatment drug | overall duration of study (5 years)
  IPF treatment drug data will be retrieved from the medical file of the participant.
The mean duration of dose reduction in days per IPF treatment drug | overall duration of study (5 years)
  IPF treatment drug data will be retrieved from the medical file of the participant.
The mean duration of drug interruption in days per IPF treatment drug | overall duration of study (5 years)
  IPF treatment drug data will be retrieved from the medical file of the participant.
The number of participants with lung transplantation | overall duration of study (5 years)
  Lung transplantation data will be retrieved from the medical file of the participant.
The (S)ADRs per IPF treatment reported which are possibly or probably related to the IPF treatment drug. | overall duration of study (5 years)
  (S)ADR data will be retrieved from the medical file of the patient.
The utilisation of health care resources by participants | overall duration of study (5 years)
  The utilisation of health care resources will be retrieved from the medical file of the patient.
The impact of IPF and IPF treatment on the severity of cough measured with the Cough-Visual Analogue Scale. | overall duration of study (5 years)
  Cough severity in the last 2 weeks was assessed at inclusion and at every follow-up visit using the Cough-VAS, a linear visual scale with 0 mm representing 'no cough' and 100 mm.
The impact of IPF and IPF treatment on quality of life measured with the SGRQ. | overall duration of study (5 years)
  The St- George's Respiratory questionnaire (SGRQ) is a 50-item questionnaire consisting of two parts. The first part evaluates the symptoms (i.e. cough, sputum production, wheezing and breathlessness) and the second part evaluates the activities (i.e. activities causing breathlessness or limited by breathlessness) and the impacts (e.g. on employment, daily life, etc.). Each question is scored as positive (i.e. =1) or negative (i.e. =0) and the total score is expressed as a percentage where 0% represents the best possible health status and 100% the worst possible health status. A total score can be obtained as well as a score for each of the three components. Data are collected at inclusion and minimal twice a year during follow-up.
The impact of IPF and IPF treatment on quality of life measured with the EQ-5D-5L questionnaire. | overall duration of study (5 years)
  The EQ-5D-5L consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels, going from no problems to extreme problems. Only 1 option can be chosen by the patient. This decision results in a 1-digit number that expresses the level selected for that dimension: no problems (=1), slight problems(=2), moderate problems(=3), severe problems(=4) and extreme problems(=5). The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where 0 mm represents 'worst health imaginable' and 100 mm representing 'best health imaginable'.
  Data are collected at Inclusion and at every follow-up visit.
The impact of IPF and IPF treatment on quality of life measured with with the K-BILD questionnaire | overall duration of study (5 years)
  Patients will receive the K-BILD questionnaire measuring their health-related quality of life. The K-BILD is a 15-item self-completed questionnaire measuring the health-related quality of life (HRQL) of patients with interstitial lung disease. It consists of three domains: breathlessness and activities, psychological and chest symptoms. Each question has a seven-point response scale resulting in a total score ranging between 0 and 100 with a higher score reflecting a higher HRQL. Data are collected at inclusion and at every follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Wim Wuyts, Phd, MD, Study Director — Universitaire Ziekenhuizen KU Leuven
Locations (9):
- Belgium (8):
  - Ziekenhuisnetwerk Antwerpen vzw, Antwerp
  - Cliniques Universitaires de Bruxelles - Hôpital Erasme, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - University Hospitals Leuven, Leuven
  - Centre Hospitalier Universitaire Sart Tilman, Liège
  - CHR de la Citadelle, Liège
  - CHU UCL Namur asbl - site Godinne, Yvoir
- Centre Hospitalier de Luxembourg (CHL)/ Luxembourg Institute of Health (LIH), Luxembourg, Luxembourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raghu G, Collard HR, Egan JJ, Martinez FJ, Behr J, Brown KK, Colby TV, Cordier JF, Flaherty KR, Lasky JA, Lynch DA, Ryu JH, Swigris JJ, Wells AU, Ancochea J, Bouros D, Carvalho C, Costabel U, Ebina M, Hansell DM, Johkoh T, Kim DS, King TE Jr, Kondoh Y, Myers J, Muller NL, Nicholson AG, Richeldi L, Selman M, Dudden RF, Griss BS, Protzko SL, Schunemann HJ; ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. Am J Respir Crit Care Med. 2011 Mar 15;183(6):788-824. doi: 10.1164/rccm.2009-040GL. PMID 21471066
- [Background] Collard HR, King TE Jr, Bartelson BB, Vourlekis JS, Schwarz MI, Brown KK. Changes in clinical and physiologic variables predict survival in idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2003 Sep 1;168(5):538-42. doi: 10.1164/rccm.200211-1311OC. Epub 2003 May 28. PMID 12773325
- [Background] Flaherty KR, Mumford JA, Murray S, Kazerooni EA, Gross BH, Colby TV, Travis WD, Flint A, Toews GB, Lynch JP 3rd, Martinez FJ. Prognostic implications of physiologic and radiographic changes in idiopathic interstitial pneumonia. Am J Respir Crit Care Med. 2003 Sep 1;168(5):543-8. doi: 10.1164/rccm.200209-1112OC. Epub 2003 May 28. PMID 12773329
- [Background] Latsi PI, du Bois RM, Nicholson AG, Colby TV, Bisirtzoglou D, Nikolakopoulou A, Veeraraghavan S, Hansell DM, Wells AU. Fibrotic idiopathic interstitial pneumonia: the prognostic value of longitudinal functional trends. Am J Respir Crit Care Med. 2003 Sep 1;168(5):531-7. doi: 10.1164/rccm.200210-1245OC. Epub 2003 Jun 5. PMID 12791580
- [Background] Fernandez Perez ER, Daniels CE, Schroeder DR, St Sauver J, Hartman TE, Bartholmai BJ, Yi ES, Ryu JH. Incidence, prevalence, and clinical course of idiopathic pulmonary fibrosis: a population-based study. Chest. 2010 Jan;137(1):129-37. doi: 10.1378/chest.09-1002. Epub 2009 Sep 11. PMID 19749005
- [Background] Marshall RP, Puddicombe A, Cookson WO, Laurent GJ. Adult familial cryptogenic fibrosing alveolitis in the United Kingdom. Thorax. 2000 Feb;55(2):143-6. doi: 10.1136/thorax.55.2.143. PMID 10639533
- [Background] Baumgartner KB, Samet JM, Stidley CA, Colby TV, Waldron JA. Cigarette smoking: a risk factor for idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 1997 Jan;155(1):242-8. doi: 10.1164/ajrccm.155.1.9001319.
- [Background] American Thoracic Society; European Respiratory Society. American Thoracic Society/European Respiratory Society International Multidisciplinary Consensus Classification of the Idiopathic Interstitial Pneumonias. This joint statement of the American Thoracic Society (ATS), and the European Respiratory Society (ERS) was adopted by the ATS board of directors, June 2001 and by the ERS Executive Committee, June 2001. Am J Respir Crit Care Med. 2002 Jan 15;165(2):277-304. doi: 10.1164/ajrccm.165.2.ats01. No abstract available. PMID 11790668
- [Background] Raghu G, Freudenberger TD, Yang S, Curtis JR, Spada C, Hayes J, Sillery JK, Pope CE 2nd, Pellegrini CA. High prevalence of abnormal acid gastro-oesophageal reflux in idiopathic pulmonary fibrosis. Eur Respir J. 2006 Jan;27(1):136-42. doi: 10.1183/09031936.06.00037005. PMID 16387946
- [Background] Meltzer EB, Noble PW. Idiopathic pulmonary fibrosis. Orphanet J Rare Dis. 2008 Mar 26;3:8. doi: 10.1186/1750-1172-3-8. PMID 18366757
- [Background] Nathan SD, Basavaraj A, Reichner C, Shlobin OA, Ahmad S, Kiernan J, Burton N, Barnett SD. Prevalence and impact of coronary artery disease in idiopathic pulmonary fibrosis. Respir Med. 2010 Jul;104(7):1035-41. doi: 10.1016/j.rmed.2010.02.008. Epub 2010 Mar 2. PMID 20199856
- [Background] Hubbard RB, Smith C, Le Jeune I, Gribbin J, Fogarty AW. The association between idiopathic pulmonary fibrosis and vascular disease: a population-based study. Am J Respir Crit Care Med. 2008 Dec 15;178(12):1257-61. doi: 10.1164/rccm.200805-725OC. Epub 2008 Aug 28. PMID 18755924
- [Background] Panos RJ, Mortenson RL, Niccoli SA, King TE Jr. Clinical deterioration in patients with idiopathic pulmonary fibrosis: causes and assessment. Am J Med. 1990 Apr;88(4):396-404. doi: 10.1016/0002-9343(90)90495-y. PMID 2183601
- [Background] Lancaster LH, Mason WR, Parnell JA, Rice TW, Loyd JE, Milstone AP, Collard HR, Malow BA. Obstructive sleep apnea is common in idiopathic pulmonary fibrosis. Chest. 2009 Sep;136(3):772-778. doi: 10.1378/chest.08-2776. Epub 2009 Jun 30. PMID 19567497
- [Background] Hubbard R, Venn A, Lewis S, Britton J. Lung cancer and cryptogenic fibrosing alveolitis. A population-based cohort study. Am J Respir Crit Care Med. 2000 Jan;161(1):5-8. doi: 10.1164/ajrccm.161.1.9906062. PMID 10619790
- [Background] Collard HR, Ryerson CJ, Corte TJ, Jenkins G, Kondoh Y, Lederer DJ, Lee JS, Maher TM, Wells AU, Antoniou KM, Behr J, Brown KK, Cottin V, Flaherty KR, Fukuoka J, Hansell DM, Johkoh T, Kaminski N, Kim DS, Kolb M, Lynch DA, Myers JL, Raghu G, Richeldi L, Taniguchi H, Martinez FJ. Acute Exacerbation of Idiopathic Pulmonary Fibrosis. An International Working Group Report. Am J Respir Crit Care Med. 2016 Aug 1;194(3):265-75. doi: 10.1164/rccm.201604-0801CI. PMID 27299520
- [Background] Martinez FJ, Safrin S, Weycker D, Starko KM, Bradford WZ, King TE Jr, Flaherty KR, Schwartz DA, Noble PW, Raghu G, Brown KK; IPF Study Group. The clinical course of patients with idiopathic pulmonary fibrosis. Ann Intern Med. 2005 Jun 21;142(12 Pt 1):963-7. doi: 10.7326/0003-4819-142-12_part_1-200506210-00005. PMID 15968010
- [Background] Gan Y, Herzog EL, Gomer RH. Pirfenidone treatment of idiopathic pulmonary fibrosis. Ther Clin Risk Manag. 2011 Feb 8;7:39-47. doi: 10.2147/TCRM.S12209. PMID 21339942